CLINICAL TRIAL: NCT05622019
Title: Evaluation of The Association Between Stage-Grade of Periodontitis and Sleep Quality and Fatigue
Brief Title: Periodontitis, Sleep Quality and Fatigue
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Tastan Eroglu, assistant professor, Necmettin Erbakan University
Other Study IDs: NecmettinEUperio
Record Dates: First submitted 2022-10-21; First posted 2022-11-18 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Periodontal Diseases; Sleep; Fatigue; Quality of Life; Healthy
Keywords: periodontal diseases; gingival health; sleep; fatigue; oral related quality of life
MeSH Terms: conditions — Periodontal Diseases; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gingival health: Healthy participants had no sites with inter-proximal attachment loss, probing pocket depth (PPD) of ≤3 mm in all sites, bleeding on probing (BOP) ≤ 10%, and had <10% of sites with modified gingival index (mGI) ≥ 2
- periodontitis: Participants were diagnosed with periodontitis if interdental clinical attachment loss (AL) was detected at ≥2 non-adjacent teeth, or buccal or oral AL was ≥3 mm with probing depth ≥3 mm was detected at ≥2 teeth.The participants in this group were divided into subgroups according to their periodontitis stage grade.

SUMMARY:
The goal of this observational study is to investigate the association of stage-grade of periodontitis with sleep quality and fatigue and the effect of periodontitis on QoL (Quality of life) in individuals with periodontitis and gingivally healthy individuals.

The main questions it aims to answer are:

1. Have poor sleep quality, inadequate sleep and fatigue got an effect on periodontal status?
2. Has periodontal status got an effect on sleep quality and fatigue?
3. What is the effect of periodontal status on quality of life?

Routine clinical and radiographic periodontal examinations of the participants were performed. Groups were designed according to periodontal status and periodontitis-stages of participants. Group 1- Healthy; Group 2- Stage I periodontitis; Group 3- Stage II periodontitis; Group 4- Stage III periodontitis; Group 5- Stage IV periodontitis. The participants were only asked to fill out the questionnaires (socio-demographic survey, tooth cleaning habit survey, The Pittsburgh Sleep Quality Index(PSQI), The Jenkins Sleep Scale(JSS), Multidimensional Assessment of Fatigue scale (MAF) and Oral Health Impact Profile-14 (OHIP-14)) included in the study and were informed about them. Then, if necessary, the participants' routine periodontal treatments were performed.

In line with the findings of the study;

1. Sleep quality was found higher in gingival healthy individuals. 3. The severity of periodontitis increases, the sleep duration becomes shorter, 4. It has been observed that the sleep quality in terms of gender is lower in female individuals compared to male individuals.

DETAILED DESCRIPTION:
This was a prospective survey study reporting on a convenience sample of 124 healthy subjects or patients with periodontitis reporting for care at the Periodontology Clinic, Necmettin Erbakan University. This study was approved by the Faculty of Dentistry Non-Pharmaceutical and Non-Medical Device Research Ethics Committee of Necmettin Erbakan University and was conducted in accordance with the Helsinki Declaration of 1975, as revised in 2013. The study participants provided a written informed consent and comprehended the assessment details fully. The investigators excluded the participants who did not comprehend the questionnaire.

Before the study, the number of patients required for each group was determined by calculating the power (G * Power 3.1 software; Heinrich Heine University, Düsseldorf, Germany). According to the power analysis results for one-way ANOVA test, the study performed on 5 groups provides 90% power and 0.37 effect size for a total of 115 samples. However, considering that there may be patients who could not continue the study, it was decided to include 124 people in the study.

Clinical measurements and stage diagnosis for all cases were performed by a single trained and calibrated investigator (KD) using Williams periodontal probes. Calibration exercise was performed in 10 non-study periodontitis patients. First, PD(probing pocket depth) and AL(attachment loss) were measured and the same protocol was repeated 1 hour later. Intra-examiner variabilities for PD and AL measurements were assessed after the completion of all measurements.

Statistical analyzes were performed with the SPSS (Statistical Package for the Social Sciences) 26.0 package program. The normality of the distribution was checked with the Kolmogorov Smirnov test. In the study, one-way anova test and Bonferroni test were used as post hoc test for comparison according to stage, grade, age and educational status, while independent sample t test was used for comparison according to gender. Pearson correlation analysis was applied to test the relationship between the scales. Chi-square analysis was used to evaluate the classification made according to sleep quality and the relationship between stage and grade. Chi-square analysis was used to evaluate the relationship between demographic characteristics and stage and grade. Statistical significance was assessed when p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age
* with no psychiatric, mental or physical disability
* those with no systemic diseases
* those with no medicine use, including antibiotics, during the previous 6 months
* without pregnancy and non-breastfeeding
* diagnosed as having healthy gingiva or periodontitis

Exclusion Criteria:

* not meet inclusion criteria
* fewer than 20 healthy teeth
* acute dental conditions that required urgent care such as an abscess, cellulitis, or diseases affecting the jawbones including cysts and neoplasms.
* history of periodontal therapy in the previous 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This was a survey study reporting on a convenience sample of 124 healty subjects or patients with periodontitis reporting for care at the Periodontology Clinic, Necmettin Erbakan University. Konya.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Investigation of the relationship between periodontitis and sleep evaluating using Pittsburgh Sleep Quality Index (PSQI) | At the beginning of the study, PSQI was applied. This process was completed within 1 month.
  The results obtained by comparing the total PSQI scores of the patients with the periodontal status of the patients constitute one of the primary results of this study.Scoring of the answers was based on a 0 to 3 scale. "5" or greater indicated a "poor" sleeper. Higher PSQI scores represented worse sleep quality.
Investigation of the relationship between periodontitis and sleep evaluating using Jenkins sleep scale(JSS) | At the beginning of the study, JSS was applied. This process was completed within 1 month. Sleep disturbances are considered when the mean score is equal or greater than 2, corresponding to at least one troubled night per week
  The results obtained by comparing the total JSS scores of the patients with the periodontal status of the patients constitute one of the primary results of this study. Sleep disturbances are considered when the mean score is equal or greater than 2, corresponding to at least one troubled night per week
Investigation of the relationship between periodontitis and fatigue | At the beginning of the study, Multidimensional Assessment of Fatigue scale (MAF) was applied. This process was completed within 1 month.
  The results obtained by comparing the total Multidimensional Assessment of Fatigue scale (MAF) scores of the patients with the periodontal status of the patients constitute one of the primary results of this study. The index score can range from 1(no fatigue) to 50 (extreme fatigue). As the score obtained from the questionnaire increases, the level of fatigue increases.
Investigation of the relationship between periodontitis and oral health related quality of life (OHrQoL) | At the beginning of the study, OHIP-14 questionnaire was applied. This process was completed within 1 month.
  OHRQoL was evaluated by using Oral Health Impact Profile-14 (OHIP-14). The results obtained by comparing the total OHIP-14 scores of the patients with the periodontal status of the patients constitute one of the primary results of this studyPatients answered their negative experiences on a 0 to 4 scale. The OHIP-14 score is the total score of the answers (0 to 56), with higher scores indicating poorer OHRQoL. Any score higher than the 14 was taken as an indication of poor OHRQoL

SECONDARY OUTCOMES:
Comparison of data with periodontal status | At the beginning of the study, Socia-demographic questionnaire was applied. This process was completed within 1 month.
  Each enrolled participant was asked to complete a questionnaire. The questionnaire consisted of the following three main parts: (i) demographic characteristics (age, educational attainment); and (ii)tooth-cleaning habits. The results of the comparison of these data with the periodontal situation constitute the secondary result of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, dentistry Faculty, Konya, Turkey (Türkiye)